CLINICAL TRIAL: NCT03685734
Title: Visual Outcomes Following Descemet Stripping Automated Endothelial Keratoplasty for Corneal Endothelial Dysfunction
Brief Title: Visual Outcomes Following Descemet Stripping Automated Endothelial Keratoplasty
Acronym: VO-DSAEK
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-13Obs-CHRMT
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Corneal Endothelial Disorder
Keywords: DSAEK

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess objective and subjective visual outcomes achieved by patients with corneal endothelial dysfunction who have undergone surgical treatment with Descemet stripping automated endothelial keratoplasty (DSAEK).

DETAILED DESCRIPTION:
Since 2006, the technique by removing the Descemet membrane from the recipient cornea was renamed Descemet stripping automated endothelial keratoplasty (DSAEK). In recent years, DSAEK techniques have evolved, favoring increasingly thinner and finer grafts, known as ultrathin DSAEK (UT DSAEK), with the aim of obtaining better visual results.

Endothelial keratoplasty is now the most common surgical procedure used to treat endothelial dysfunction. The current study focused on assessing both objective and subjective visual quality outcomes following DSAEK.

ELIGIBILITY:
Inclusion Criteria:

* Clinical eligibility for DSAEK
* Informed written consent
* Successful completion of DSAEK procedure
* Postoperative follow-up at least 1 year
* Ability to respond to the questionnaire

Exclusion Criteria:

* Patients with clinical edematous cornea
* With significant stromal opacity
* With major disturbances of ocular surface
* Previous corneal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with corneal endothelial dysfunction underwent DSAEK
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  Scored with reference to the logarithm of the minimum angle of resolution (logMAR) and its variation in line gain.